CLINICAL TRIAL: NCT05717582
Title: A Prospective Study of Maximal-Cytoreductive Therapies for Patients With de Novo Metastatic Hormone-sensitive Prostate Cancer Who Achieve Oligopersistent Metastases During Systemic Treatment With Apalutamide Plus ADT (CHAMPION Study)
Brief Title: Maximal Cytoreductive Therapies on Post-treatment Metastases in Pts With mHSPC During Apalutamide Plus ADT Treatment
Acronym: CHAMPION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCa-CHAMPION
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Prostate Cancer; Castration-Sensitive Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maximal-cytoreductive therapy (Experimental): Patients with de novo mCSPC who achieve ≤10 oligopersistent metastases on PSMA PET CT after initial 3-month systemic treatment with apalutamide plus ADT will receive cytoreductive radical prostatectomy with/without PLND and metastasis-directed therapy with radiation.
  Interventions: Drug: apalutamide; Drug: androgen deprivation therapy; Procedure: cytoreductive radical prostatectomy with/without pelvic lymph node dissection; Radiation: metastasis-directed therapy with radiation

INTERVENTIONS:
Drug: apalutamide — Patients receive apalutamide 240mg,qd,po.
Drug: androgen deprivation therapy — Patients receive systemic ADT.
Procedure: cytoreductive radical prostatectomy with/without pelvic lymph node dissection — Patients receive cytoreductive radical prostatectomy with/without pelvic lymph node dissection.
Radiation: metastasis-directed therapy with radiation — Patients receive metastasis-directed therapy with radiation guided by post-treatment oligopersistent metastases.

SUMMARY:
To assess the feasibility and safety of Maximal cytoreductive therapies in patients with de novo mCSPC who achieve ≤10 oligopersistent metastases on PSMA PET CT after initial 3-month systemic treatment with apalutamide plus ADT. Maximal cytoreductive therapies consist of 1.cytoreductive radical prostatectomy with/without PLND guided by post-treatment PET 2.metastasis-directed therapy with radiation guided by post-treatment oligopersistent metastases. All patients receive continuous systemic treatment with apalutamide plus ADT.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the informed consent;
2. Aged ≥18 years;
3. Histologically or cytologically confirmed prostate adenocarcinoma (primary small cell carcinoma or signet-ring cell carcinoma of the prostate are not allowed, however adenocarcinoma with neuroendocrine differentiation accounting ≤10% is allowed);
4. Newly diagnosed prostate cancer (within 3 months prior to enrollment);
5. M1a/b disease with the presence of 1-10 visible metastases at diagnosis by conventional imagine including bone scan (ECT) and CT or MRI of the chest, abdomen, and pelvis;
6. With initial systemic treatment of apalutamide plus ADT and willing and expected to comply with treatment and follow up schedule [No more than 2-month systemic treatment before enrollment (including ADT and ADT combined with short-term first-generation anti-androgen therapy (flutamide or bicalutamide); To maximize enrollment, patients who had started apalutamide plus ADT before enrollment are allowed into the study provided that they are otherwise eligible and therapy was initiated no longer than 2 months before enrollment];
7. Fit to undergo cytoreductive radical prostatectomy and radiotherapy to the visible sites of metastases;
8. ECOG PS score is 0-1;
9. Adequate organ function;
10. Life expectancy ≥ 12 months.

Exclusion Criteria:

1. History of allergies, hypersensitivity, or intolerance to any drug used in the study;
2. Had the contraindications or is intolerant to cRP or RT;
3. Had any visceral metastases (brain, liver, lung etc.) on screening conventional imaging (bone scans, CT or MRI);
4. Prior Received any of the following treatments for primary and metastatic prostate cancer;

   1. >2-month ADT or first-generation antiandrogens (bicalutamide, flutamide etc.);
   2. Any other novel hormonal therapies (enzalutamide, darolutamide, abiraterone etc.) except ≤ 2-month apalutamide plus ADT listed in inclusion criteria;
   3. Any chemotherapy;
   4. local treatment or metastatic treatment for primary prostate cancer or metastases;
   5. Any immunotherapy (PD-L1 etc.), target therapy (PARPi etc), etc;
5. History of seizure or known condition that may predispose to seizure;
6. History of major surgery 4 weeks before enrollment;
7. Had major cardiovascular and cerebrovascular diseases within 6 months prior to the start of the study;
8. Any condition that could interfere with drug absorption(e.g. unable to swallow, chronic diarrhea etc. );
9. Conditions of active infection;
10. History of previous or current malignant disease, except for curatively treated tumors cured for more than 3 years;
11. Patients who is currently undergoing other trials;
12. Unwilling or difficult to cooperate with treatment and follow-up visit;
13. Other sever conditions which could interfere with trial safety or results judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with undetectable PSA level after 6 cycles of treatment (each cycle is 28 days). | At the end of the 6th cycle of treatment (each cycle is 28 days).
  It is defined as the proportion of patients with PSA≤0.2 ng/mL without disease progression or symptomatic deterioration after 6 cycles of study treatment (each cycle is 28 days).

SECONDARY OUTCOMES:
proportion of patients with undetectable PSA level after 3 cycles of treatment (each cycle is 28 days). | At the end of the 3rd cycle of treatment (each cycle is 28 days).
  It is defined as the proportion of patients with PSA≤0.2 ng/mL after 3 cycles of study treatment (each cycle is 28 days).
PSA50 response rate and PSA90 response rate at the end of the 3rd treatment cycle (each cycle is 28 days). | At the end of the 3rd cycle of treatment (each cycle is 28 days).
  It is defined as the proportion of patients with a PSA reduction of over 50% / 90%compared with baseline.
PSA50 response rate and PSA90 response rate at the end of the 6th treatment cycle (each cycle is 28 days). | At the end of the 6th cycle of treatment (each cycle is 28 days).
  It is defined as the proportion of patients with a PSA reduction of over 50% / 90%compared with baseline.
Conventional imaging and PSMA-PET/CT imaging features at baseline | Baseline (Before trial treatment)
  Imaging features before hormonal therapy
Proportion of patients with ≤ 10 metastases on PSMA-PET/CT imaging at the end of the third treatment cycle (each cycle is 28 days). | At the end of the 3rd cycle of treatment (each cycle is 28 days).
  Proportion of patients with ≤ 10 metastases on PSMA-PET/CT imaging at the end of the third treatment cycle (each cycle is 28 days).
Comparison of imaging features between conventional imaging and PSMA PET/CT. | At the end of the 3rd and 6th cycle of treatment (each cycle is 28 days).
  Including prostate volume, tumor burden, distribution of metastatic lesions etc.
Feasibility and safety of performing cRP±MDT treatment | At the end of the 6th cycle of treatment (each cycle is 28 days).
  Feasibility and safety of performing cRP±MDT guided by oligopersistent metastases assessed by PSMA PET/CT

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center Pudong Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center Xuhui Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Wang B, Pan J, Zhang T, Ni X, Wei Y, Li X, Fang B, Hu X, Gan H, Wu J, Wang H, Ye D, Zhu Y. Protocol for CHAMPION study: a prospective study of maximal-cytoreductive therapies for patients with de novo metastatic hormone-sensitive prostate cancer who achieve oligopersistent metastases during systemic treatment with apalutamide plus androgen deprivation therapy. BMC Cancer. 2024 May 25;24(1):643. doi: 10.1186/s12885-024-12395-3. PMID 38796422